CLINICAL TRIAL: NCT01233024
Title: Satiety Response of Fructo-oligosaccharide (FOS), Inulin, Soluble Corn Fiber (SCF), and Resistant Starch (RS) in Overweight Woman and Relationship to Fermentation
Brief Title: Satiety Response of Four Dietary Fibers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 1003E78714
Record Dates: First submitted 2010-05-28; First posted 2010-11-02 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: Adult; Women; Dietary Fiber; Satiety Response; Food Intake
MeSH Terms: interventions — Resistant Starch; fructooligosaccharide; Inulin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Low fiber control (Placebo Comparator): no treatment dinner bar, no treatment breakfast bar
  Interventions: Dietary Supplement: Control
- Promitor soluble corn fiber (Experimental): 12g in dinner bar, 11g in breakfast bar
  Interventions: Dietary Supplement: Soluble corn fiber
- FiberSym resistant starch (Experimental): 12g in dinner bar, 11g breakfast bar
  Interventions: Dietary Supplement: Resistant starch
- Orafti P95 fructooligosaccharide (Experimental): 12g in dinner bar, 11g in breakfast bar
  Interventions: Dietary Supplement: Fructooligosaccharide
- Orafti HPX inulin (Experimental): 12g in dinner bar, 11g in breakfast bar
  Interventions: Dietary Supplement: Inulin

INTERVENTIONS:
Dietary Supplement: Control — Dinner bar fortified with 0g fiber; breakfast bar fortified with 0g dietary fiber.
  Other Names: Low fiber control
  Arms: Low fiber control
Dietary Supplement: Soluble corn fiber — Dinner bar fortified with 12g fiber; breakfast bar fortified with 11g dietary fiber.
  Other Names: Promitor soluble corn fiber
  Arms: Promitor soluble corn fiber
Dietary Supplement: Resistant starch — Dinner bar fortified with 12g fiber; breakfast bar fortified with 11g dietary fiber.
  Other Names: FiberSym resistant starch
  Arms: FiberSym resistant starch
Dietary Supplement: Fructooligosaccharide — Dinner bar fortified with 12g fiber; breakfast bar fortified with 11g dietary fiber.
  Other Names: Orafti P95 fructooligosaccharide
  Arms: Orafti P95 fructooligosaccharide
Dietary Supplement: Inulin — Dinner bar fortified with 12g fiber; breakfast bar fortified with 11g dietary fiber.
  Other Names: Orafti HPX inulin
  Arms: Orafti HPX inulin

SUMMARY:
Studies have found a relationship between dietary fiber consumption and body weight regulation. This relationship may stem from enhanced satiety through fermentation of certain fibers in the large intestine.

The objective of this study is to determine and compare satiety ratings, changes in food intake, and gastrointestinal effects for four fibers: fructooligosaccharide, inulin, soluble corn fiber, and resistant starch.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* Age 18-40 years
* Nonsmoking
* Not taking weight loss medications
* Non-dieting (weight has not changed more than 11 pounds over three months)
* BMI between 18.5 and 29
* Spoken and written English literacy

Exclusion Criteria:

* Do not regularly consume breakfast
* Food allergies to wheat, soy, peanut, or dairy
* BMI less than 25 or greater than 29 upon admission to study
* Cancer diagnosis in past 5 years
* History of heart disease, kidney disease, diabetes, or eating disorder
* History of ulcerative colitis, Crohn's disease, or any other gastrointestinal condition
* History of drug or alcohol abuse in past 6 months
* Use of lipid-lowering, anti-hypertensive, or anti-inflammatory steroid medication
* Concurrent or recent (within 30 days) intervention study participation
* Pregnant or lactating
* Irregular menstrual cycle
* Vegetarians
* People who eat more than approximately 15 grams of fiber per day

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Satiety response using visual analogue scales | 0, 15, 30, 45, 60, 90, 120, 180 minutes postprandially
  Satiety response will be measured using subjective perceptions of hunger, fullness, satisfaction, and prospective food intake evaluated by previously validated visual analogue scales (VAS).

SECONDARY OUTCOMES:
Food intake | 180 minutes postprandially and over 24 hours
Breath hydrogen response | 0 and 180 minutes
Gastrointestinal tolerance using visual analogue scales (VAS) | 24 hours
  Subjective ratings of bloating, stool consistency, and flatulence will be measured using VAS. A stool count will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne L Slavin, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Saint Paul, Minnesota, United States